CLINICAL TRIAL: NCT07089940
Title: An Early Phase 1 Trial to Assess Pharmacodynamic Effects of OMO-103 in Patients With Pancreatic Ductal Adenocarcinoma
Brief Title: OMO-103 for the Treatment of Locally Advanced or Metastatic Pancreatic Ductal Adenocarcinoma
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00027995; NCI-2025-05087 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00027995 (Other: OHSU Knight Cancer Institute); P30CA069533 (NIH)
Record Dates: First submitted 2025-07-22; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Locally Advanced Pancreatic Ductal Adenocarcinoma; Metastatic Pancreatic Ductal Adenocarcinoma; Stage II Pancreatic Cancer AJCC v8; Stage III Pancreatic Cancer AJCC v8; Stage IV Pancreatic Cancer AJCC v8
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (OMO-103) (Experimental): Patients receive OMO-103 IV over 30-45 minutes on days 1 and 8 in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI, tumor biopsies, and collection of blood samples throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Myc Inhibitor OMO-103

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Myc Inhibitor OMO-103 — Given IV
  Other Names: OMO 103; OMO-103; OMO103

SUMMARY:
This early phase I trial studies the biological activity of OMO-103 in patients with pancreatic ductal adenocarcinoma that has spread to nearby tissue or lymph nodes (locally advanced) or that has spread from where it first started (primary site) to other places in the body (metastatic). OMO-103 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. This trial may help researchers determine how exposure to OMO-103 changes pancreatic tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the pharmacodynamic effects of Myc inhibitor OMO-103 (OMO-103) in tumor biopsies from patients with pancreatic ductal adenocarcinoma (PDAC).

SECONDARY OBJECTIVE:

I. To assess safety and tolerability of the proposed therapy.

EXPLORATORY OBJECTIVE:

I. To identify predictive biomarkers of sensitivity to therapy.

OUTLINE:

Patients receive OMO-103 intravenously (IV) over 30-45 minutes on days 1 and 8 in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) or magnetic resonance imaging (MRI), tumor biopsies, and collection of blood samples throughout the study.

After completion of study treatment, patients are followed up at 30 days and then for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Must provide written informed consent before any study-specific procedures or interventions are performed
* Must be ≥ 18 years old at the time of informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Clinically-confirmed diagnosis of locally-advanced or metastatic adenocarcinoma of the pancreas

  * Participants may be treatment naïve or have received prior therapy for the treatment of their PDAC. A minimum washout period of 14-days after completing the most recent line of therapy is required before a participant can initiate treatment with study agent(s)
* Based on available imaging, participant must have at least one disease lesion that can be biopsied in accordance with institutional standards
* Patient agrees to undergo a minimum of 2 biopsies (pre- and post-treatment). Note: at principal investigator (PI) discretion, archival sample may be obtained in lieu of pre-treatment biopsy
* Hemoglobin ≥ 7.5 g/dL
* Absolute neutrophil count (ANC) ≥ 1.0 x 10^9/L (> 1500 per mm^3)
* Platelet count ≥ 75 x 10^9/L (> 100,000 per mm^3)
* Calculated creatinine clearance > 50 mL/min/1.73m^2 (per Cockcroft-Gault equation)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT): ≤ 3 x upper limit of normal (ULN), or ≤ 5 x ULN in presence of liver metastases
* Participants of childbearing potential (POCBP) must agree to abstain from sexual intercourse or use effective methods of contraception starting with the first dose of study therapy through 6 months from the last dose of study intervention
* POCBP may participate provided they have a negative serum pregnancy test at screening and a negative serum OR urine pregnancy test within 7 days of starting treatment
* Sperm-producing participants must agree to abstain from sexual intercourse or use effective contraception starting with the first dose through 6 months after last dose of study intervention

Exclusion Criteria:

* Concomitant use of other anti-cancer therapy otherwise not permitted in this protocol, including: chemotherapy, immunotherapy, hormonal therapy (hormone replacement therapy is acceptable), radiotherapy (except for palliative), biological therapy, or other novel agent
* Prior anti-cancer therapy within 2 weeks prior to study enrollment
* Prior treatment with a MYC inhibitor
* Known severe hypersensitivity to OMO-103 or to any excipient of these medicinal products, or history of allergic reactions attributed to compounds of similar chemical or biologic composition
* Major surgery within 6 weeks prior to enrollment
* Uncontrolled intercurrent illness including symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, and myocardial infarction within 3 months of initiating study intervention
* History of psychiatric illness likely to interfere with ability to comply with protocol requirements or give informed consent
* Participant is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 6 months after the last dose of trial treatment
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Measurable change in tumor biology | Time of pretreatment biopsy (baseline) to completion of post-treatment biopsy
  A change in tumor biology is defined as any difference in the cellular or molecular composition of the tumor or its surrounding environment that can be quantifiably measured between the pre- and post-treatment tissue samples. Will be reported as a binary outcome of observed change (e.g., yes/no) for each participant.

SECONDARY OUTCOMES:
Incidence of treatment-related adverse events | Day 1 (i.e., start of study intervention) up to 30 days after last dose of study drug
  Will be assessed according to Common Terminology Criteria for Adverse Events version 5.0. The exact 95% confidence interval will be reported with the point estimate of toxicity rate.

CONTACTS AND LOCATIONS:
Overall Officials: Charles D Lopez, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States